CLINICAL TRIAL: NCT01848886
Title: Endoscopic Versus Open Radial Artery Harvest and Mammario-radial Versus Aorto-radial Grafting in Patients Undergoing Coronary Artery Bypass Surgery (The 2x2 Factorial Designed Randomised NEO Trial)
Brief Title: Neurological Complications Comparing Endoscopically vs. Open Harvest of the Radial Artery
Acronym: NEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Christian Lildal Carranza, MD, Head of Adult Cardiac Surgery, Executive-MBA, Rigshospitalet, Denmark
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: H-3-2012-116; H-3-2012-116 (Other: Ethics Committee)
Record Dates: First submitted 2013-02-25; First posted 2013-05-08 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Complications Due to Coronary Artery Bypass Graft; Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases
Keywords: ERAH; Endoscopic Radial Artery Harvest; Y-graft; Radial Artery Harvest; Total Arterial Revascularisation; CABG; Radial Artery Conduit
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Grp 1: ERAH, Mammarioradial (Y-graft) (Other): Endoscopic radial artery harvest Mammarioradial graft (Y-graft) In this group the radial artery is harvested as an endoscopic procedure and positioned on the heart as an composite graft (Y-graft).
  Interventions: Procedure: Endoscopic radial artery harvest; Procedure: Mammarioradial graft (Y-graft)
- Grp 2: ERAH, Aortoradial (Free RA) (Other): Endoscopic radial artery harvest Aortooradial (free RA) In this group the radial artery is harvested as an endoscopic procedure and positioned on the heart as an free RA graft.
  Interventions: Procedure: Endoscopic radial artery harvest; Procedure: Aortoradial graft (Free RA)
- Grp 3: ORAH, Mammarioradial (Y-graft) (Other): Open radial artery harvest Mammarioradial graft (Y-graft) In this group the radial artery is harvested as an open procedure and positioned on the heart as an composite graft (Y-graft).
  Interventions: Procedure: Open radial artery harvest; Procedure: Mammarioradial graft (Y-graft)
- Grp 4: ORAH, Aortoradial graft (Free RA) (Other): Aortooradial graft (free RA) Open radial artery harvest In this group the radial artery is harvested as an open procedure and positioned on the heart as an free RA graft.
  Interventions: Procedure: Open radial artery harvest; Procedure: Aortoradial graft (Free RA)

INTERVENTIONS:
Procedure: Endoscopic radial artery harvest — Radial artery harvest is performed as an endoscopic procedure.
  Arms: Grp 1: ERAH, Mammarioradial (Y-graft); Grp 2: ERAH, Aortoradial (Free RA)
Procedure: Open radial artery harvest — Radial artery harvest is performed as an open procedure.
  Arms: Grp 3: ORAH, Mammarioradial (Y-graft); Grp 4: ORAH, Aortoradial graft (Free RA)
Procedure: Mammarioradial graft (Y-graft) — The radial artery is used as an composite graft positioned on the internal mammarian artery.
  Arms: Grp 1: ERAH, Mammarioradial (Y-graft); Grp 3: ORAH, Mammarioradial (Y-graft)
Procedure: Aortoradial graft (Free RA) — The radial artery is used as an free graft positioned on the aorta.
  Arms: Grp 2: ERAH, Aortoradial (Free RA); Grp 4: ORAH, Aortoradial graft (Free RA)

SUMMARY:
Coronary artery bypass grafting (CABG) using the radial artery (RA) has since the nineties gone through a revival. The initially reported worse outcome in RA graft patients compared to patients grafted with the saphenous vein (SV) has since been corrected. Studies have shown better patency when using RA, so the RA is going to be preferred more and more especially in younger patients where long time patency is critical. During the last 10 years endoscopic techniques to harvest the RA have evolved. Multiple different techniques have been used, but now the equipment and technique have been refined and are highly reliable. The investigators hypothesize that the endoscopic technique has less complications and a just as good patency as open harvest. There are also two possible ways to use the RA as a graft. One way is sewing it onto the aorta and another way is sewing it onto the mammarian artery. The investigators hypothesize that using it on the mammarian artery is superior as a revascularisation technique with just as good a patency as sewing it directly onto the aorta.

DETAILED DESCRIPTION:
Objectives

The present trial will in patients undergoing CABG (1) evaluate the complications in endoscopic versus traditionally harvested radial arteries, (2) evaluate graft patency in endoscopic harvested radial arteries versus open technique, and (3) evaluate the use of mammario-radial grafting versus aorto-radial grafting.

Design and trial size

The NEO Trial is a randomised clinical trial with a 2x2 factorial design. We plan to randomise 300 participants into four intervention groups: (1) mammario-radial endovascular group; (2) aorto-radial endovascular group; (3) mammario-radial open group and (4) aorto-radial open group. A subgroup of 100 participants will be selected to undergo a special scanning of the vascular perfusion of donor and control hands (MIBI scan). The evaluation of graft patency and ischaemia in the arm will be blinded but the assessment of the primary outcome of handfunction at three months is non-blinded evaluated by questionnaire.

Trial interventions

Trial 1: The experimental procedure in this trial will be endoscopic radial artery harvest (ERAH). The control intervention will be open radial artery harvest (ORAH).

Trial 2: The experimental procedure in this trial will be the technique where the radial artery is sewn onto the mammarian artery as a mammario-radial anastomosis (composite/Y-graft). The control intervention will be the technique of sewing the radial artery directly onto the aorta as an aorto-radial anastomosis (free radial artery).

Inclusion and exclusion criteria

All patients referred to our department for sub acute or elective coronary bypass operation will be eligible for trial inclusion. Inclusion criteria are: 18 years or older; able and willing to give informed consent; multi-vessel disease. Exclusion criteria are: off-pump procedure; multi-procedure (i.e. concomitant valve surgery); contrast allergy; geographically not available for follow-up; Allen's test with insufficient ulnary artery perfusion; no informed consent; acute operation; dialysis; preoperative neurological deficit on the donor arm; left ventricle ejection fraction (LVEF) less than 20%; former sternotomy and malignant disease.

Primary and secondary outcomes

Trial 1: The primary outcome will be evaluation of hand function at three months.

The secondary outcomes will be: occurrence of neurophysiological defects in the donor arm assessed by examination of cutaneous sensibility and measurements of the sensory and motoric nervous conduction velocity preoperatively and after three months; change in subjective cutaneous sensibility assessed by a clinical examination after three months; complications assessed as a composite of haematoma formation, wound dehiscence or infection registered before discharge and after three months.

We will also assess a number of exploratory outcomes (serious adverse events, reoperation for bleeding, revascularisation, myocardial infarction, stroke or death, handgrip strength, muscular function in the hand, scar evaluation, vascular supply to the hand, graft patency and participants subjective evaluation of hand function after 1 year).

Trial 2: The primary outcome will be the occurrence of cardio- or cerebrovascular events during the first year after surgery comparing mammario-radial versus aorto-radial grafts. As an exploratory outcome we will also assess graft patency by multi-slice computer tomography (MSCT) comparing mammarioradial versus aortoradial grafts one year after surgery.

Time schedule

Randomisation will commence after 15th of May 2013. The inclusion period of altogether 300 participants is expected to last three years.

ELIGIBILITY:
Inclusion Criteria

* Elective/sub acute CABG as an isolated procedure.
* Age > 18 years
* Multi-vessel disease
* Non-dominant arm is eligible for radial artery harvest
* Written informed consent

Exclusion Criteria

* Geographically not available for follow up
* Modified Allen's test indicating insufficient ulnary artery perfusion
* Valve surgery, ablation surgery or any kind of concomitant surgery during same admission.
* Acute operation (<24 hours from admission)
* Dialysis
* Preoperative neurological deficit on the donor arm
* LVEF < 20% preoperative
* Former sternotomy
* Contrast allergy
* Malignant disease
* No written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2013-05; Primary Completion 2018-10 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Sum score of hand function questionnaire | 3 months postoperatively
  Using Likert-type scale scoring system quality of life is assessed after radial artery harvest. The mean values in the ERAH group will be compared to the mean value in the ORAH group at three months after surgery.
Occurence of cardiac and cerebrovascular events in aortoradial versus mammarioradial grafting | 1 year postoperatively
  Occurrence of one of the following cardiac or cerebrovascular events: all cause mortality, myocardial infarction (MI), target vessel revascularisation (TVR) or stroke at one year postoperatively will be compared.

SECONDARY OUTCOMES:
Complications in the donor arm in ERAH versus ORAH | 3 months postoperatively
  Occurrence of complications at three months after surgery. Complications are defined as a composite of haematoma formation, wound dehiscence, or infection will be compared.
Clinical neurological examination in donor arm ERAH versus ORAH | 3 months postoperatively
  Clinical examination of subjective cutaneous sensibility will be compared between ERAH versus ORAH groups.
Neurological deficits in ERAH versus ORAH | 3 months postoperatively
  Occurence of deficits in following neurological exams will be compared between ERAH and ORAH
  1. Cutaneous sensibility on both forearms and hands by appraisal of dermatomes. All sensibility modalities are examined:
     1. Cutaneous touch sensibility examined by Von Fray hair
     2. Deep pain sensibility examined by algometry.
  2. Sensory nervous conduction velocity examined on both forearms and hands:
     1. N. medianus (dig. II - hdl); orthodromic technique
     2. N. ulnaris (dig. V - hdl); orthodromic technique
     3. N. radialis (antebrachium - tabatiere); antidromic technique
     4. N. cutaneous antebrachium lateralis (elbow - antebrachium); antidromic technique
     5. N. cutaneous antebrachium medialis (elbow - antebrachium); antidromic technique
  3. Motoric nervous conduction velocity examined on both forearms and hands:
     1. N. medianus (hdl - m. abductor policis brevis (APB), elbow - APB)
     2. N. ulnaris (hdl - m. abductor digiti minimi)

OTHER OUTCOMES:
Vascular function in the donor arm of the ERAH and ORAH groups compared to non-donor arms. | 3 months postoperatively
  MIBI scan after exercise induced relative ischemia will be compared between donor versus non-donor arms.
Graft patency in ERAH versus ORAH | 1 year postoperatively
  MSCT will be used to evaluate patency.
Graft patency in aortoradial versus mammarioradial grafting | 1 year postoperatively
  MSCT will be used to evaluate patency.
Change in handgrip strength | the day before surgery and 1 year postoperatively.
  Change in handgrip strength will be measured in the conduit donor arm and compared between ERAH versus ORAH.
Change in muscular function in ERAH versus ORAH | the day before surgery and 1 year postoperatively
  Following muscles are rated according to the Oxford Scale for grading muscle strength (see table 7) the day before surgery and at one year postoperatively:
  * m. abductor pollicis brevis
  * m. abductor digiti minimi
  * mm. interosseus palmares
  * m. flexor digitorum profundus II+V
  * m. extensor digitorum The change in muscular function will be compared between ERAH versus ORAH.
Serious adverse events in ERAH versus ORAH | 1 year postoperatively
  Occurrence of the following serious adverse events at time point one year after surgery: reoperation for bleeding; revascularisation; myocardial infarction; stroke; or death will be compared between ERAH and ORAH.
Scar evaluation in ERAH versus ORAH | 1 year postoperatively
  Using Stony Brooke Scar Evaluation Score the scars will be evaluated and the mean scores compared between ERAH versus ORAH groups.
Neuropathic pain symptoms and signs in ERAH versus ORAH | 3 months postoperatively
  The Leeds assessment of neuropathic symptoms and signs (LANNS) pain scale will be used after 3 months to compare pain in ERAH versus ORAH groups.

CONTACTS AND LOCATIONS:
Overall Officials: Christian L Carranza, MD, Principal Investigator — Department of Cardio-Thoracic Surgery, Rigshospitalet, Copenhagen, Denmark; Peter Skov Olsen, MD DMSc, Study Chair — Department of Cardio-Thoracic Surgery, Rigshospitalet, Copenhagen, Denmark; Christian Gluud, MD DMSc, Study Chair — Copenhagen Trial Unit, Rigshospitalet, Copenhagen, Denmark; Martin Ballegaard, MD PhD, Study Chair — Department of Clinical Neurophysiology, Rigshospitalet, Copenhagen, Denmark; Philip Hasbak, MD PhD, Study Chair — Department of Clinical Physiology, Nuclear Medicine and PET, Rigshospitalet, Copenhagen, Denmark; Andreas Kjær, Prof MD DMSc, Study Chair — Department of Clinical Physiology, Nuclear Medicine and PET, Rigshospitalet, Copenhagen, Denmark; Klaus F Kofoed, MD DMSc, Study Chair — Department of Cardiology and Radiology, Rigshospitalet, Copenhagen, Denmark; Mads Werner, MD, DMSc, Study Chair — Multidisciplinary Pain Centre, Rigshospitalet, Copenhagen, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Carranza CL, Petersen JJ, Ballegaard M, Werner MU, Hasbak P, Kjaer A, Kofoed KF, Lindschou J, Gluud C, Olsen MH, Engstrom J, Jakobsen JC. Endoscopic or Open Radial Artery Harvest in Coronary Artery Bypass Surgery. NEJM Evid. 2026 Jan;5(1):EVIDoa2500199. doi: 10.1056/EVIDoa2500199. Epub 2025 Dec 23. PMID 41432491
- [Derived] Carranza CL, Ballegaard M, Werner MU, Hasbak P, Kjaer A, Kofoed K, Olsen MH, Gluud C, Jakobsen JC. Detailed statistical analysis plan for the neurological complications in endoscopic versus open radial artery harvest (NEO) randomised clinical trial. Trials. 2022 Dec 9;23(1):990. doi: 10.1186/s13063-022-06869-7. PMID 36494849
- [Derived] Carranza CL, Ballegaard M, Werner MU, Hasbak P, Kjaer A, Kofoed KF, Lindschou J, Jakobsen JC, Gluud C, Olsen PS, Steinbruchel DA. Endoscopic versus open radial artery harvest and mammario-radial versus aorto-radial grafting in patients undergoing coronary artery bypass surgery: protocol for the 2 x 2 factorial designed randomised NEO trial. Trials. 2014 Apr 23;15:135. doi: 10.1186/1745-6215-15-135. PMID 24754891